CLINICAL TRIAL: NCT00360464
Title: A Multicenter, Non-Randomized, Open Label Trial Of Azithromycin SR For The Treatment Of Acute Bronchitis And Secondary Infection Of Chronic Respiratory Diseases In Japan Adults
Brief Title: A Trial Of Azithromycin SR For The Treatment Of Acute Bronchitis And Secondary Infection Of Chronic Respiratory Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661175
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

INTERVENTIONS:
Drug: Azithromycin SR

SUMMARY:
To evaluate the clinical efficacy and safety in patients with Acute Bronchitis or Secondary Infection of Chronic Respiratory Diseases receiving a dose of 2 g of azithromycin in the SR formulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as mild or moderate in severity by the classification of infection of the Japanese Society of Chemotherapy guidelines for the evaluation methods of new antibacterial drug (established in 1997).

Exclusion Criteria:

* Severe underlying disease; patients in which drug clinical evaluation is difficult because of confounding diseases.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is investigator's clinical efficacy at Day 8.

SECONDARY OUTCOMES:
Endpoints of efficacy are as follows: Investigator's clinical efficacy (at Day 15 and 29), and the tendency toward clinical improvement (at Day 4); Bacteriological efficacy (at Day 4, 8, 15 and 29); Safety Endpoints: Adverse events and safety lab data.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Japan (18):
  - Pfizer Investigational Site, Hitachi-Naka, Ibaraki
  - Pfizer Investigational Site, Kasama, Ibaraki
  - Pfizer Investigational Site, Moriya, Ibaraki
  - Pfizer Investigational Site, Toride, Ibaraki
  - Pfizer Investigational Site, Tsuchiura, Ibaraki
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Yokosuka, Kangawa
  - Pfizer Investigational Site, Kami-gun, Miyagi
  - Pfizer Investigational Site, Shigesato-cho, Nagasaki, Nagasaki
  - Pfizer Investigational Site, Shindoori, Niigata-shi, Niigata
  - Pfizer Investigational Site, Katano, Osaka
  - Pfizer Investigational Site, Akiruno, Tokyo
  - Pfizer Investigational Site, Chōfu, Tokyo
  - Pfizer Investigational Site, Kodaira, Tokyo
  - Pfizer Investigational Site, Nakano City, Tokyo
  - Pfizer Investigational Site, Setagaya City, Tokyo
  - Pfizer Investigational Site, Shinagawa, Tokyo
  - Pfizer Investigational Site, Yonezawa, Yamagata

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661175&StudyName=A%20Trial%20Of%20Azithromycin%20SR%20For%20The%20Treatment%20Of%20Acute%20Bronchitis%20And%20Secondary%20Infection%20Of%20Chronic%20Respiratory%20Diseases